CLINICAL TRIAL: NCT04309188
Title: Effect of Stroboscopic Vision Training in a Softball Season: A Randomized Controlled Trial Pilot Study
Brief Title: Stroboscopic Vision Training in Softball
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L20-095
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Sports Performance; Vision, Ocular
Keywords: Stroboscopic; Vision Training; Softball; On-field performance

STUDY DESIGN:
Intervention Model Description: The pilot study will use a pre-test post-test randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Vision Center and balance assessor will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroboscopic Training Group (Experimental): Treatment group, which will receive stroboscopic training during hitting and fielding drills. The glasses look like sunglasses but have liquid crystal technology that causes a flicker from clear to opaque. The glasses flickering will be controlled on the side of the glasses by the researcher. When the athlete can complete a skill proficiently by catching or hitting during training the level of flickering will be increased to challenge the visual system more.
  Interventions: Device: Senaptec Strobe Glasses
- Standard softball drills (Active Comparator): Control group, which will perform normal hitting and fielding drills without stroboscopic training
  Interventions: Other: Standard softball drills

INTERVENTIONS:
Device: Senaptec Strobe Glasses — The glasses use liquid crystal technology that causes a flicker from clear to opaque to enhance vision.
  Arms: Stroboscopic Training Group
Other: Standard softball drills — Control group, which will perform normal hitting and fielding drills without stroboscopic training
  Arms: Standard softball drills

SUMMARY:
Enhanced sports performance, in our current world, is being pushed at the professional level and down to school-age children as well. Money is being spent on lessons and equipment to enhance performance. One new method to enhance performance is stroboscopic vision goggles. The glasses lenses flicker removing visual information for a brief moment. The claim is that they train connections between the eyes, brain, and body. We want to see if this product truly does enhance visual performance during a softball season for high school girls.

DETAILED DESCRIPTION:
In today's sports world, every strategy to perform at the highest level is needed. Current literature is demonstrating enhanced sports performance using stroboscopic vision training.1,2,5 The objective of this randomized controlled trial is to measure the effect of a stroboscopic visual training in a high school softball season in comparison to controls. Athletes in the control group will go through normal practice drills for hitting and fielding. The stroboscopic training (experimental group) will use the strobe glasses during hitting and fielding drills two times a week in practice. The brand of strobe glasses is Senaptec Strobe. Athletes in both the experimental and control groups will have their vision assessed at the beginning of the season and end by The West Texas Vision Center. Measurements for vision will include developmental eye movement, vergence ranges, Randot stereopsis test, accommodative ranges, acuity, and stereo scores. On-field performance measurements will be collected for batting statistics including on-base percentage, batting average, slugging percentage, and hard-hit ball percentage in both the experimental and control groups. The current year batting statistics will be compared with the prior year statistics if enough at-bats occurred. In addition, to the vision and on-field hitting performance proprioception balance using the Balance Error Scoring System (BESS) will be measured at the beginning of the season and end for both groups. Our data will provide quantified information for coaches, athletes, and health care providers concerning the benefits of the strobe glasses warrant buying to enhance sports performance. Additionally, we wish to determine whether visual-motor and proprioception balance changes occur after the training.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 14-18 years 2) females; 3) high school softball

Exclusion Criteria:

* 1) Prior use of stroboscopic vision training; 2) History of seizures; 3) History of vestibular impairments

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Results are needed for softball that only females play in high school.
Enrollment: 34 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Vergence ranges | 8 weeks
  Vergence ranges measured how many prism diopters the subject can turn their eyes in (base out) and how far they can relax them out (base in). This score is also a good measure of how much peripheral fusion a person has.

SECONDARY OUTCOMES:
Developmental eye movement | 8 weeks
  Developmental eye movement will measure how fast the subject can track numbers vertically and horizontally.
Randot stereopsis test | 8 weeks
  Randot stereopsis test will measures how many ARC seconds of stereo the subject has. This test measures the subject's magno and parvocellular stereo tracking their peripheral or central fusion.
Accommodative ranges | 8 weeks
  Accommodative ranges will measure how many times the subject can clear an image looking through a plus and minus accommodation flipper in thirty seconds.
Acuity | 8 weeks
  Acuity will measure the clarity of vision at a distance of twenty feet.
Stereo Scores | 8 weeks
  Stereo Scores will measure how quickly the athlete recognizes depth perception
Batting statistics | 8 weeks
  Batting statistics including on-base percentage, batting average, slugging percentage, hard-hit ball percentage will be provided by the coach at the end of the season for the current year and prior year. Subjects will need a minimum of 20 at-bats in a season for collection of these statistics.
Balance Error Scoring System (BESS) | 8 weeks
  Balance Error Scoring System (BESS) measures the total number of postural errors committed in a 30-second trial standing on flat surface and foam pad. It provides a measure of balance and proprioceptive ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appelbaum LG, Cain MS, Schroeder JE, Darling EF, Mitroff SR. Stroboscopic visual training improves information encoding in short-term memory. Atten Percept Psychophys. 2012 Nov;74(8):1681-91. doi: 10.3758/s13414-012-0344-6. PMID 22810559
- [Background] Ballester R, Huertas F, Uji M, Bennett SJ. Stroboscopic vision and sustained attention during coincidence-anticipation. Sci Rep. 2017 Dec 20;7(1):17898. doi: 10.1038/s41598-017-18092-5. PMID 29263340
- [Background] Mitroff SR, Friesen P, Bennett D, Yoo H, Reichow AW. Enhancing ice hockey: Skills through stroboscopic visual training: A Pilot Study. Athl Train Sports Health Care. 2013;5(6):261-264
- [Background] Wilkins L, Nelson C, Tweddle S. Stroboscopic visual training: A pilot study with three elite youth football goalkeepers. J Cogn Enhanc. 2018;2:3-11.
- [Background] Hays JB, Korba BE. DNA from recombinogenic lambda bacteriophages generated by arl mutant of Escherichia coli is cleaved by single-strand-specific endonuclease S1. Proc Natl Acad Sci U S A. 1979 Dec;76(12):6066-70. doi: 10.1073/pnas.76.12.6066. PMID 160560 (Retraction: PMID 3883350 Hays JB, Korba BE. Proc Natl Acad Sci U S A. 1985 Feb;82(3):953)
- [Background] Grooms DR, Chaudhari A, Page SJ, Nichols-Larsen DS, Onate JA. Visual-Motor Control of Drop Landing After Anterior Cruciate Ligament Reconstruction. J Athl Train. 2018 May;53(5):486-496. doi: 10.4085/1062-6050-178-16. Epub 2018 May 11. PMID 29749751